CLINICAL TRIAL: NCT02591043
Title: Surgical Treatment of Low Energy Pelvic Ring Fractures in the Elderly: Cross-sectional Single-centre Study From Basel, Switzerland
Brief Title: Surgical Treatment of Low Energy Pelvic Fractures in the Elderly
Acronym: PelvicRetro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-299
Record Dates: First submitted 2015-10-08; First posted 2015-10-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Fracture
Keywords: Pelvic; Treatment Outcome
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Follow-up (Other): Patients have not received a structured follow up examination or evaluation of outcome after surgery. Therefore this study aims at conducting a follow up examination regarding functional outcome, pain and radiologic healing in these patients.
  Interventions: Procedure: Outcome after surgery

INTERVENTIONS:
Procedure: Outcome after surgery — Functional outcome after surgical treatment of pelvic ring fractures Measurements: TUG-test score, ADLs index, maximal pain (VAS 1-10) at rest and experienced during TUG-test. One-year mortality, signs of healing, dislocation or other complications on anterior-posterior radiographs of the pelvis, living situation before and after the injury (at home/institutional placement)

SUMMARY:
Since May 2010 the Department of Trauma, Basel University Hospital has performed surgical stabilisation of the posterior pelvic ring on 55 patients. These patients have not received a structured follow up examination or evaluation of outcome after surgery.

DETAILED DESCRIPTION:
Functional outcome of elderly patients with surgical treatment of low energy pelvic ring fractures.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age ≥55y ears) of any ethnic / sociodemographic background
* Pelvic ring fracture after low energy trauma affecting the posterior ring or both (posterior and anterior ring)
* Surgical stabilisation of the pelvic ring at Basel University Hospital between May 2010 and December 2014
* Ambulatory before surgery
* Informed consent for study participation by the patient or legal representatives

Exclusion Criteria:

* Refusal of consent by the patient or legal representatives to participate in the study
* Fractures within the last 3 months before follow-up
* Suspicion of a pathological fracture in the context of known or unknown malignancy
* Symptomatic low back pain with morphological changes, i.e. intervertebral disc displacement, neoplasm metastasis in the axial skeleton, spinal stenosis, vertebral fracture, spondylarthropathy etc.
* Pre-trauma mobility status that precludes achieving a post-trauma mobility status enabling the patient to perform the timed up and go test (e.g. patient in a wheel chair)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
TUG-Test through study completion, an average of 1 year | through study completion, an average of 1 year
  TUG test - according test description

SECONDARY OUTCOMES:
activity of daily living (ADL) through study completion, an average of 1 year | through study completion, an average of 1 year
  ADL test - according test description
Pain test through study completion, an average of 1 year | through study completion, an average of 1 year
  Maximal pain (VAS 1-10) experienced during TUG-test and at rest at the day of follow up
Living Situation through study completion, an average of 1 year | through study completion, an average of 1 year
  Living situation before and after the injury (at home/institutional placement) according test procedure
1-year mortality | one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hasler, Dr, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Rommens PM, Hofmann A. Comprehensive classification of fragility fractures of the pelvic ring: Recommendations for surgical treatment. Injury. 2013 Dec;44(12):1733-44. doi: 10.1016/j.injury.2013.06.023. Epub 2013 Jul 18. PMID 23871193